CLINICAL TRIAL: NCT06225310
Title: A Phase I Trial of Selinexor, Ruxolitinib and Methylprednisolone for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Trial of Selinexor, Ruxolitinib and Methylprednisolone
Acronym: KPT-IST-391
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPT-IST-391
Record Dates: First submitted 2023-11-07; First posted 2024-01-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; Multiple Myeloma, Refractory; Multiple Myeloma in Relapse
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; ruxolitinib; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Selinexor/Ruxolitinib/Steroids (Other): The regimen will follow a 3+3 dose escalation schedule starting at dose level 0. Subjects enrolled at dose level 0 will receive 1) selinexor (once weekly) starting at 40 mg, 2) ruxolitinib (twice a day (BID) on days 1-28) starting at 10 mg, and 3) oral methylprednisolone (every other day (QOD)) a set dose at 40 mg. Subjects at dose level 1 will receive 1) selinexor (once weekly) 60 mg, 2) ruxolitinib (BID) on days 1-28 10 mg, and 3) methylprednisolone (QOD) 40 mg. Subjects at dose level 2 will receive 1) selinexor (once weekly) 60 mg, 2) ruxolitinib (BID) on days 1-28 15 mg, and 3) oral methylprednisolone (QOD) 40 mg.
  Interventions: Drug: Selinexor; Drug: Ruxolitinib; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Selinexor — Selinexor (KPT-330) is a first-in-class, oral selective exportin 1 (XPO1) inhibitor (1,2). Selinexor functions by binding with and inhibiting the nuclear export protein XPO1 (also called CRM1), leading to the accumulation of tumor suppressor proteins in t
  Other Names: XPOVIO
Drug: Ruxolitinib — elective inhibitor of Janus kinase (JAK)
  Other Names: Jakafi
Drug: Methylprednisolone — Glucocorticoid, steroid
  Other Names: Medrol

SUMMARY:
Selinexor, a first-in-class, oral selective exportin 1 (XPO1) inhibitor, has shown promise in pre-clinical and clinical studies. It functions by inhibiting the nuclear export protein XPO1, resulting in the accumulation of tumor suppressor proteins and inhibition of oncoprotein mRNAs, which is selectively lethal to myeloma cells. Selinexor has demonstrated activity in combination with various drugs, including glucocorticoids and proteasome inhibitors, leading to its FDA approval for the treatment of relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Selinexor, a first-in-class, oral selective exportin 1 (XPO1) inhibitor, has shown promise in pre-clinical and clinical studies. It functions by inhibiting the nuclear export protein XPO1, resulting in the accumulation of tumor suppressor proteins and inhibition of oncoprotein mRNAs, which is selectively lethal to myeloma cells. Selinexor has demonstrated activity in combination with various drugs, including glucocorticoids and proteasome inhibitors, leading to its FDA approval for the treatment of relapsed or refractory multiple myeloma.

Ruxolitinib, an oral JAK1/2 inhibitor, has been approved by the FDA for myelofibrosis treatment. Preliminary experiments have shown that Ruxolitinib, in combination with lenalidomide and dexamethasone, effectively inhibits MM cell proliferation. Additionally, the combination of Ruxolitinib and dexamethasone has demonstrated enhanced anti-MM effects. Clinical results indicate that Ruxolitinib in combination with steroids is well-tolerated in heavily treated MM patients.

This proposed study aims to investigate the efficacy of a lower dose of Selinexor in combination with Ruxolitinib and methylprednisolone for patients with relapsed/refractory multiple myeloma. The study builds on the existing evidence of the individual and synergistic effects of Selinexor and Ruxolitinib, both in preclinical and clinical settings and seeks to provide a potential new treatment option for MM patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible to enroll in this study:

1. Has a diagnosis of MM based on standard criteria as follows:

Myeloma criteria: Must be At least 1 of 2 1. Clonal bone marrow plasma cells >10% 2. Biopsy-proven bony or extramedullary plasmacytoma

Active Myeloma criteria: Active Myeloma criteria: Must Meet At Least ONE of the Following:

Meet at least one of the sub-criteria for #1 Evidence of End Organ Damage (a, b, c, or d), OR Meet sub-criteria #2. 60% or greater bone marrow plasma cells, OR Meet sub-criteria #3 Serum free light chain ratio, OR Meet sub-criteria #4 More than one focal lesion on MRI > 5mm in size.

1. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically

   1. Hypercalcemia: serum calcium >0.25 mmol/L (>1mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11mg/dL)
   2. Renal insufficiency: creatinine clearance <40 mL per minute or serum creatinine >177mol/L (>2mg/dL)
   3. Anemia: hemoglobin value of >20g/L below the lowest limit of normal, or a hemoglobin value <100g/L
   4. Bone lesions: one or more osteolytic lesion on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
2. 60% or greater clonal plasma cells on bone marrow examination
3. Serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100 mg/L (a patient's involved free light chain either kappa or lambda is the one that is above the normal reference range; the uninvolved free light chain is the one that is typically in, or below, the normal range)
4. More than one focal lesion on MRI that is at least 5mm or greater in size

The patient must have met the criteria for Active Myeloma at some stage following the diagnosis of Myeloma. Source documentation for both Myeloma and Active Myeloma will be required.

2. Patients with relapsed/refractory multiple myeloma with at least three prior lines of therapy 3. Received an

1. Anti-CD38 antibody
2. Immunomodulatory agent (IMiD)
3. Proteasome inhibitor (PI) 4. Currently has MM with measurable disease, defined as:

   * a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or urine monoclonal protein levels of at least 200 mg/24 hours
   * for patients without measurable serum and urine M-protein levels, an involved SFLC > 100 mg/L or abnormal SFLC ratio
   * for patients with IgD MM, a monoclonal immunoglobulin IgD of at least 5500 mg/L or meet other measurable disease eligibility criteria
   * for patients with IgA MM, total IgA of > 700 mg/dL 5. Currently has progressive MM: MM patients that are relapsed or have refractory disease from at least 3 regimens or lines of therapy are eligible for enrollment provided they fulfill the other eligibility criteria:
   * patients are considered relapsed, when they progress greater than 60 days from their last dose of treatment
   * patients are refractory when they progress while currently receiving the treatment or within 8 weeks of its last dose 6. Adequate hepatic function within 14 days prior to C1D1: Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to < 2 × ULN.

     7. Adequate renal function within 14 days prior to C1D1 as determined by OR estimated CrCl of > 60 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female (87)(Appendix 5).

     8. Adequate hematopoietic function within 14 days prior to C1D1: total WBC count ≥1500/mm3, ANC ≥1000/mm3, hemoglobin ≥8.5 g/dL and platelet count ≥75,000/mm3 (patients for whom <50% of BM nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of BM nucleated cells are plasma cells).

     9. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, G-CSF, GM-CSF, and platelet stimulators (e.g., eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.

     10. Patients must have:
   * At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the start of study treatment
   * At least a 1-week interval from the last platelet transfusion prior to the start of study treatment
   * However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study 11. Female patients of childbearing potential (FCBP) must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active must use highly effective methods of contraception throughout the study and for one month following the last dose of study treatment. Male patients must agree not to donate sperm during the study treatment period. Specifically:
   * FCBP† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting treatment and must either commit to continued abstinence from heterosexual intercourse or use acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts therapy. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

     † A FCBP (female of childbearing potential) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) 12. Able to take antiplatelet therapy if platelet count is above 30 x 109/L. Options include aspirin (acetylsalicylic acid, ASA) at 81 or 325/mg/daily, warfarin low molecular weight hepairin, Pradaza, Eliquis, or Xarelto.

     13. Patients with history of human immunodeficiency virus (HIV) are eligible if they have CD4+ T cell counts ≥350 cells/µL, negative viral load per institutional standard, and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year.

     14. Patients with untreated hepatitis C virus (HCV) are eligible if there is a documentation of negative viral load per institutional standard.

     15. Age ≥ 18 years of age. 16. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.

     17. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

1. Patients who had prior exposure to ruxolitinib or selinexor
2. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) during the 3 years prior to randomization. Cancer treated with curative intent for >5 years previously and without evidence of recurrence will be allowed.
3. Have light chain amyloidosis
4. Have plasma cell leukemia
5. Have history of active tuberculosis
6. Have any concurrent medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, POEMS syndrome [polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes], primary amyloidosis, etc.) that is likely to interfere with study procedures.
7. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
8. Received the following prior therapy:

   * Chemotherapy within 3 weeks of study drugs
   * Corticosteroids (>20 mg/daily prednisone or equivalent) within 3 weeks of study drugs to ensure that steroid dose intensity at the beginning of the treatment is not altered by administration of steroids prior to the study. Consumption of steroids within 3 weeks of the treatment may interfere with efficacy and side effects due to differences of steroid intensity.
   * Immunotherapy, immunomodulatory drugs, or proteasome inhibitors within 3 weeks before administration of study drugs
   * Extensive radiation therapy within 28 days before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
   * Use of any other experimental drug or therapy within 28 days of study drugs
   * Strong CYP3A4 inhibitors, strong CYP3A4 inducers and fluconazole doses >200 mg daily within 5 half-lives before study drugs. (For example, clarithromycin has half-life of 4 hours so washout period for clarithromycin is 20 hours.)
9. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
10. Known hypersensitivity to compounds of similar chemical or biological composition to ruxolitinib or steroids.
11. Concurrent use of other anti-cancer agents or treatments.
12. Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin
13. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
14. Pregnant or breastfeeding females.
15. Body surface area (BSA) <1.4 m2 at baseline, calculated by the Dubois or Mosteller method.
16. Life expectancy of less than 3 months.
17. Major surgery within 4 weeks prior to C1D1.
18. Active, unstable cardiovascular function, as indicated by the presence of:

    1. Symptomatic ischemia, or
    2. Uncontrolled clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on anti-arrhythmic are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
    3. CHF of New York Heart Association Class ≥3 or known left ventricular ejection fraction < 40%, or
    4. Myocardial infarction (MI) within 3 months prior to C1D1 or
    5. Stroke and other thrombosis, such as, pulmonary embolism (PE) or deep vein thrombosis (DVT) within 3 months prior to C1D1.
19. Any active GI dysfunction interfering with the patient's ability to swallow tablets, or any active GI dysfunction that could interfere with absorption of study treatment.
20. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Comprehensive Cancer Network® (NCCN) Clinical Practice Guidelines in Oncology (CPGO) (NCCN CPGO) for antiemesis and anorexia/cachexia (palliative care).
21. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
22. Contraindication to any of the required concomitant drugs or supportive treatments.
23. Patients unwilling or unable to comply with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
1. Maximum Tolerated Dose (MTD): | 30 months
  ● A standard 3 + 3 dose escalation schedule will be used for all escalations
2. Recommended phase 2 dose (RP2D) | 30 months
  Primary objective of a phase 1 study is to define a safe and tolerable dose to use in further studies designed to determine efficacy, the Recommended Phase 2 Dose (RP2D)

SECONDARY OUTCOMES:
1. Overall Response Rate ([ORR]=CR+VGPR+PR) | 30 months
  ORR is a measure of how many patients in a study experience a significant reduction or complete disappearance of their cancer following treatment, essentially indicating the percentage of patients who have a partial or complete response to the therapy being tested. ORR is calculated by adding the number of patients with a "Complete Response" + Very Good Partial Response + Partial Response.
2. Clinical Benefit Rate ([CBR]=CR+VGPR+PR+MR) | 30 months
  The percentage of patients with advanced cancer who experience a complete or partial response to a treatment. CBR is calculated by adding the number of patients with Complete Response (CR) + Very Good Partial Response (VGPR) + Partial Response (PR) + Minor Response.
3. To determine disease parameters for study treatment: | 30 months
  * Time to progression (TTP) - define as the time from the initiation of therapy to progressive disease
  * Progression-free survival (PFS) - defined as the time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
  * Time to first response - defined as the time from the initiation of therapy to the first evidence of confirmed clinical benefit defined as > minimal response (MR, including patients who achieved a complete response (CR), very good partial response (VGPR), partial response (PR), or MR
  * DOR - defined as the time from the first response to progressive disease
  * Overall survival (OS) - Overall survival, defined as the time from initiation of therapy to death from any cause or last follow-up visit

OTHER OUTCOMES:
Background and rationale for assessment of serum B cell maturation antigen levels (sBCMA) | 30 months
  Only for MM patients participating in the optional biomarker including sBCMA analysis study.
  To evaluate the ability of MM-related biomarkers including sBCMA, to serve as:
  * Diagnostic biomarker by determining specificity and sensitivity in MM patients
  * Prognostic biomarker by determining its ability to predict the probable course of the disease including its recurrence.
  * Stratification biomarker by examining its ability to predict clinical outcomes of MM patients

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (1):
- Berenson Cancer Center, West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No